CLINICAL TRIAL: NCT02393521
Title: The Effect of Vibration Therapy on Pressure Pain Thresholds Over Neck Myofascial Trigger Points: a Randomized Controlled Study
Brief Title: The Effect of Vibration Therapy Over Neck Myofascial Trigger Points
Acronym: vibraMTrP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Lirios Dueñas, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1421077978677
Record Dates: First submitted 2015-02-22; First posted 2015-03-19 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Myofascial Trigger Point Pain; Neck Pain
Keywords: Vibration; Pressure Pain Threshold; Trigger Points; Neck Pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vibration group (Experimental): Patients in the vibration therapy group received 10 self-administered sessions of vibration therapy (45-50 Hz), one session per day, remaining on their Shindo® vibration mattress at home in supine for 15 min.
  Interventions: Device: Shindo® vibration mattress
- Control group (No Intervention): Subjects in the control group did not receive vibration therapy

INTERVENTIONS:
Device: Shindo® vibration mattress — vibration therapy was self-administered while the subject was laying in supine in a polyurethane mattress
  Other Names: vibration therapy
  Arms: Vibration group

SUMMARY:
The aim of this study was to investigate the efficacy of a self-administered vibration therapy treatment on neck pain, disability and pressure pain thresholds in patients with non-specific neck pain and myofascial trigger points (MTrPs). The investigators hypothesized that patients receiving vibration therapy would report less perceived neck pain, disability and present higher PPTs after receiving vibration therapy when compared to a control no-treatment group.

DETAILED DESCRIPTION:
Myofascial trigger points (MTrPs) are a common source of (regional) pain in patients presenting with musculoskeletal pain. Mechanical vibration has been suggested as a treatment for pain relief. In this study, the effects of vibration therapy on people with non-specific neck pain and MTrPs were investigated. Seventeen chronic non-specific neck pain patients were randomly assigned to a treatment (vibration group, n = 9) or control group (n = 8). Vibration group received 10 self-administered sessions of vibration therapy (45-50 Hz for 15 minutes with the subject laying in supine). Perceived neck pain and disability and pressure pain thresholds over MTrPs of the upper trapezius and levator scapulae bilateraly were measured at baseline and after the first, five and 10 treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* a score of ≥ 5/50 in Neck Disability Index
* active or latent myofascial trigger points in upper trapezius or levator scapulae muscles

Exclusion Criteria:

* previous cervical spine surgery
* cervical radiculopathy
* severe systemic disease
* fibromyalgia
* other widespread musculoskeletal pain syndromes
* patients being treated with medication or physiotherapy within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | 10 days
  Pain tolerance was measured at baseline (T0) and after the first (T1), five (T5) and 10 treatment sessions (T10).

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | 10 days
  Perceived neck pain and disability were measured at baseline (T0) and after the first (T1), five (T5) and 10 treatment sessions (T10).

CONTACTS AND LOCATIONS:
Overall Officials: Sofía Pérez, PhD, Study Director — University of Valencia
Locations (1):
- Universitat de Valencia, Valencia, Spain

REFERENCES:
- [Result] Imtiyaz S, Veqar Z, Shareef MY. To Compare the Effect of Vibration Therapy and Massage in Prevention of Delayed Onset Muscle Soreness (DOMS). J Clin Diagn Res. 2014 Jan;8(1):133-6. doi: 10.7860/JCDR/2014/7294.3971. Epub 2014 Jan 12. PMID 24596744